CLINICAL TRIAL: NCT03894826
Title: A Phase 2 Clinical Trial Testing the Safety and Efficacy of Voronistat in Pediatric Patients With Drug Resistant Epilepsy
Brief Title: Voronistat in Pediatric Patients With Drug Resistant Epilepsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VOR-17-2471
Record Dates: First submitted 2018-09-13; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Refractory Epilepsy
Keywords: PEDIATRIC
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TREATMENT (Experimental): Participants will be administered 230 mg/m2/day of oral Vorinostat [100 mg tablets] in addition to standard of care anti-seizure medication for a duration of 6 weeks.
  Interventions: Drug: Vorinostat 100 MG

INTERVENTIONS:
Drug: Vorinostat 100 MG — Vorinostat administered by mouth, once daily at a dose of 230 mg/m2/day for a total of 6 weeks
  Other Names: ZOLINZA

SUMMARY:
The study evaluates the safety, tolerability, and efficacy of Vorinostat in addition to standard of care anti-epileptic drugs in pediatric patients with medically refractory epilepsy. All participants entering the treatment phase will receive Vorinostat.

DETAILED DESCRIPTION:
Vorinostat is a potent inhibitor of histone deacetylases (HDAC). HDACs catalyze the removal of acetyl groups from the lysine residues of proteins, including histones and transcription factors. Valproic acid, a broad anti-epileptic drug, commonly used as first line treatment in epilepsy, has also been shown to inhibit HDAC activity .

It is it is anticipated that Vorinostat in a population of pediatric patients with epilepsy will be well-tolerated, similar to that seen with valproic acid and other normally prescribed anti-epileptic drugs.

Participants consenting to participate will enter a 4-week screening period to ensure eligibility. Eligible participants will then enter the 6-week treatment phase. Participants will be seen for a final Safety Follow-up visit 6 weeks after end of treatment. Participants who are enrolled and complete all study procedures will be in the study for a total of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 2 - 17 years (inclusive)
2. Medically intractable epilepsy, defined as having failed at least 2 standard anti-seizures therapies and experiencing at least 3 motor seizures per week, separated by at least 24 hours that are quantifiable by observation (e.g. discrete episodes of motor activity). Participants experiencing other seizure types in addition to motor seizures may also be enrolled but must meet the minimal requirement for motor seizures.
3. Ability and willingness of family and/or caregiver (when appropriate) to give written informed consent and to comply with requirement of the study
4. Adequate bone marrow function (defined as an absolute neutrophil count (ANC) of > 2 x 109/L; platelet count of > 150 x 109/L; hemoglobin of > 110 g/L [3-11 years], > 120 g/L [females 12 years or over], > 125 g/L [males 12-14 years], > 137 g/L [males 15 years or older])
5. Adequate renal function (defined as serum creatinine < 1.5X age-adjusted upper limit of normal [ULN], or glomerular filtration rate ≥ 70 mL/min/1.73 m2)
6. Adequate hepatic function (defined as total bilirubin <1.5 times ULN, and alanine aminotransferase [ALT] and aspartate transaminase [AST] < 3 times ULN, and albumin >33 g/L)
7. Corrected QT (QTc) interval of < 450 msec
8. Prothrombin time (PTT) < 1.5 ULN/International Normalized Ratio (INR) < 1.5 ULN
9. Participants on corticosteroids must be taking a stable or decreasing dose for at least 7 days prior to enrollment

Exclusion Criteria:

1. Treatment with valproic acid or other HDACi class drugs within at least the last 3 months at time of screening
2. Enzyme-inducing AEDs (including oxcarbazepine (Trileptal), phenobarbital, phenytoin (Dilantin), topiramate (Topamax)
3. Coumarin-derivative anti-coagulants
4. Participants being considered for surgery for management of seizures during screening or who will be receiving surgery during for management of seizures during study period (includes all neurosurgery for the management of seizures or device implantation for the management of seizures)
5. Neurosurgery within the past 12 months
6. Use of Vagus Nerve Stimulator (VNS) where settings have not been stable for at least 6 months
7. Planned surgery or other invasive medical treatment during screening of during treatment period
8. Hypokalemia or hypomagnesemia
9. Participants starting or currently on any neurometabolic diet (including but not limited to ketogenic diet; medium-chain triglyceride diet; modified Atkins diet; low glycemic index diet) during study
10. History of non-catheter related deep venous thrombosis
11. Pleural effusion
12. Malignancy within the past 5 years.
13. Any serious medical condition that according to the investigator could interfere with the conduct of the study
14. Serious comorbid disease in which the life expectancy of the patient is shorter than the duration of the trial
15. Unwillingness or inability to comply with study requirements
16. Positive pregnancy test, lactating females or heterosexually active participants not willing to use highly effective methods of contraception
17. Participation in any clinical trial with an investigational drug, or therapy not approved by Health Canada, within one month prior to screening

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 14 days post drug initiation; 30 days post drug initiation; 42 days post drug initiation; 42 days following drug discontinuation
  The number of treatment emergent adverse events will be tabulated at each time point: adverse events, serious adverse events, and discontinuations due to adverse events.
Incidence of Drug Discontinuations due to Adverse Drug Reaction | 14 days post drug initiation; 30 days post drug initiation; 42 days post drug initiation; 42 days following drug discontinuation
  The number of participants with drug discontinuations due to Adverse Drug Reaction will be tabulated at each time point: adverse events, serious adverse events, and discontinuations due to adverse events.

SECONDARY OUTCOMES:
Proportion of participants who have at least a 50% reduction in seizures from baseline | 42 days post drug initiation; change from baseline
  Treatment response will be evaluated by calculating the proportion of response of participants who demonstrate a 50% reduction rate or greater at 6 weeks as compared to baseline.
Change in seizure status at each time point. | 14 days post drug initiation; 30 days post drug initiation; 42 days post drug initiation; 42 days following drug discontinuation
  Seizure status will be tabulated 14 days following drug initiation; 30 days following drug initiation; 42 days following drug initiation; and 42 days following drug discontinuation. Seizure status will be defined as: significant response (at least 50% reduction in seizure frequency as compared to baseline, or no seizures while on medication; partial response (25% - 49% reduction in seizure frequency as compared to baseline); no change, (0 - 24% reduction in seizure frequency as compared to baseline); and worsening (increase in seizure frequency as compared to baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Jong Rho, MD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Result] Ibhazehiebo K, Gavrilovici C, de la Hoz CL, Ma SC, Rehak R, Kaushik G, Meza Santoscoy PL, Scott L, Nath N, Kim DY, Rho JM, Kurrasch DM. A novel metabolism-based phenotypic drug discovery platform in zebrafish uncovers HDACs 1 and 3 as a potential combined anti-seizure drug target. Brain. 2018 Mar 1;141(3):744-761. doi: 10.1093/brain/awx364. PMID 29373639
- [Derived] Garcia AA, Koperniku A, Ferreira JCB, Mochly-Rosen D. Treatment strategies for glucose-6-phosphate dehydrogenase deficiency: past and future perspectives. Trends Pharmacol Sci. 2021 Oct;42(10):829-844. doi: 10.1016/j.tips.2021.07.002. Epub 2021 Aug 10. PMID 34389161

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT03894826/Prot_SAP_000.pdf